CLINICAL TRIAL: NCT02083471
Title: Cow's Milk and Hen's Egg Hyposensitization in Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UTU-ClinAll-0112
Record Dates: First submitted 2014-03-05; First posted 2014-03-11 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Egg Allergy; Cow's Milk Allergy
MeSH Terms: conditions — Egg Hypersensitivity; Milk Hypersensitivity | interventions — Eggs; Milk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SOTI (Active Comparator): Specific Oral Tolerance Induction with Egg or Cow's milk
  Interventions: Dietary Supplement: Specific Oral Tolerance Induction with Egg or Cow's milk
- Food Allergy follow-up (No Intervention)

INTERVENTIONS:
Dietary Supplement: Specific Oral Tolerance Induction with Egg or Cow's milk
  Arms: SOTI

SUMMARY:
Egg, milk and cereal allergies are the most important food allergies in Finnish children, the prevalence in western countries is 1-4 %. In some individuals food-allergy is maintained in to adulthood. Recent studies suggest that specific oral tolerance induction (SOTI) provides a treatment option in children with continuing allergy with high success rates. The study aims at specific oral tolerance induction in adults allergic to cow's milk or hen's egg. Oral immunotherapy involves taking very small amounts of the allergen, and slowly increasing the amount. Consequently, an elimination diet may be wholly or partially cancelled, without the fear of serious allergic reactions. Another aim is to explore changes in antibody-mediated and cell-mediated immune response to individual components of cow's milk and egg allergens during tolerance induction and compare these with the effect of the treatment.

DETAILED DESCRIPTION:
Background

Egg, milk and cereal allergies are the most important food allergies in Finnish children, the prevalence in western countries is 1-4 %. In some individuals food-allergy is maintained in to adulthood. The mainstay of treatment of IgE-mediated milk and egg allergy is an avoidance diet and carrying an epinephrine injector in case of an allergic reaction. Avoidance diet is very difficult and has negative effects on quality of life. Accidentally having milk or egg can cause life-threatening reactions, even lead to death. Recent studies suggest that specific oral tolerance induction (SOTI) provides a treatment option in children with continuing allergy with high success rates.

It is obvious that oral immunotherapy has impact on the milk and egg specific immune responses, but the mechanisms of this treatment have been studied only little and its effects on the cell and molecular level is practically unknown. There neither are any laboratory studies to monitor the efficacy or predict the outcome in advance or at the early stages of treatment. No research data is available on the humoral IgE, IgG4 and Immunoglobulin A (IgA) responses or the cell-mediated or cytokine responses induced by the individual major cow's milk and egg allergen components during oral immunotherapy. No tools exist for forecasting the outcome of the treatment.

Aims

The study aims at specific oral tolerance induction in adults allergic to cow's milk or hen's egg. Oral immunotherapy involves taking very small amounts of the allergen, and slowly increasing the amount. Consequently, an elimination diet may be wholly or partially cancelled, without the fear of serious allergic reactions. Another aim is to explore changes in antibody-mediated and cell-mediated immune response to individual components of cow's milk and egg allergens during tolerance induction and compare these with the effect of the treatment.

Materials and methods

The study will recruit 40 adult patients with either milk or egg allergy. Eligibility criteria are: 1) adults over 16 years, 2) elevated serum levels of specific IgE (≥ 5 kU/l, (kilounit per liter) milk or egg) or a positive skin-prick- test (≥ 5 mm, milk or egg), and 3) a positive milk- or egg-challenge. The recruited subjects meeting entry criteria are randomized to a tolerance induction group receiving milk or egg (n = 20) or to a control group to be followed on an avoidance diet (n = 20). Oral immunotherapy involves initially taking a very small amount of the allergen, and slowly increasing the amount gradually until a maintenance dose is reached. Up-dosing is monitored in hospital. Thereafter, the patient will continue the daily use of milk or egg at home.

Skin-prick-tests with milk or egg specific allergen components are performed, a symptom questionnaire is filled and blood samples are taken before commencement of the study, when the maintenance dose is reached and after 12 months from initiation of the study. Patient visits are carried out in outpatient clinic as part of the normal routine.

Commercially available (Thermo Fisher Scientific Phadia) specific allergen components are examined (IgE and IgG4), as well as IgA, IgA1 and IgA2. Cow's milk allergen components are: alfa-lactalbumin, beta-lactoglobulin, casein, lactoferrin and bovine serum albumin, and egg allergen components are: ovomucoid, ovalbumin, conalbumin and lysozyme.

Mononuclear leukocytes are isolated from the blood samples and cultured in 37 ° C incubator 10^6 cells per millilitre of RPMI (Roswell Park Memorial Institute Medium) medium containing 5% autologous plasma and cows' milk allergen components: alfa-lactalbumin, beta-lactoglobulin, bovine serum albumin, casein and lactoferrin, or egg allergen components: ovomucoid, ovalbumin, conalbumin and lysozyme. Mitogen is used as the positive control and medium without stimulation as the negative control. Milk and egg allergen components are cleaned with Detoxi-Gel Endotoxin Removal Gel columns (Thermo Scientific Pierce Chemicals) to remove effects of endotoxins during cell stimulation. Lymphoproliferation is studied using three parallel samples and cytokine expression is studied using two parallel samples (Luminex/Lincoplex: interleukin-4 (IL-4), IL-5, IL-10, IL-12, IL-13, IL-17, IL-18, IL-22, IL-23, IL-27, interferon gamma(IFN-γ), tumor necrosis factor (TNF) and transforming growth factor beta (TGF-β)).

Ethical considerations

Study follows instructions and regulations used in biomedical research. The Turku University Ethics committee approved the study 15th February 2011. Each participant will give written informed consent. Research participation is voluntary and may be suspended without any reason at any time during the study and the refusal or termination shall not affect the patient's other treatment. Patient samples and the data collected are processed and stored according to the instructions and regulations used in biomedical research.

Estimate, schedule and results

Patient visits are carried out in outpatient clinics as part of the normal reception of allergy patients and do not entail additional costs to the patients. The expenses related to antibody-mediated and cell-mediated immune response studies are covered by external funding. The study will begin in autumn 2014 and aims being completed in the spring of 2016. The results will be published in international scientific journals.

ELIGIBILITY:
Inclusion Criteria:

* Allergy to Egg or Cow's milk verified by challenge history and specific IgE

Exclusion Criteria:

* Cardiovascular disease
* Active immunological disease

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with negative results | 12 months after commencement

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Savolainen, MD Professor, Principal Investigator — University of Turku